CLINICAL TRIAL: NCT05852691
Title: A Phase II, Multicenter, Randomized, Double-Blind Study of Tobemstomig/RO7247669 Combined With Nab-Paclitaxel Compared With Pembrolizumab Combined With Nab-Paclitaxel in Participants With Previously Untreated, PD-L1-Positive, Locally-Advanced Unresectable or Metastatic Triple-Negative Breast Cancer
Brief Title: A Study of Tobemstomig + Nab-Paclitaxel Compared With Pembrolizumab + Nab-Paclitaxel in Participants With Previously Untreated, PD-L1-Positive, Locally-Advanced Unresectable or Metastatic Triple-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CO44194
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants will receive tobemstomig every 3 weeks, plus nab-paclitaxel administered on a repeating schedule of 3 weeks on, 1 week off, until disease progression or until up to 24 months after the first treatment, whichever is sooner.
  Interventions: Drug: Tobemstomig; Drug: Nab-Paclitaxel
- Arm B (Active Comparator): Participants will receive pembrolizumab every 3 weeks, plus nab-paclitaxel administered on a repeating schedule of 3 weeks on, 1 week off, until disease progression or until up to 24 months after the first treatment, whichever is sooner.
  Interventions: Drug: Pembrolizumab; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Tobemstomig — Participants will receive intravenous (IV) tobemstomig every 3 weeks (Q3W) until disease progression or until up to 24 months after the first treatment, whichever is sooner.
  Other Names: RO7247669
  Arms: Arm A
Drug: Pembrolizumab — Participants will receive IV pembrolizumab Q3W until disease progression or until up to 24 months after the first treatment, whichever is sooner.
  Arms: Arm B
Drug: Nab-Paclitaxel — Participants will receive IV nab-paclitaxel weekly for 3 weeks, followed by 1 week off, until disease progression or until up to 24 months after the first treatment, whichever is sooner.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of a novel immunotherapy candidate, tobemstomig, in combination with nab-paclitaxel, for patients with previously untreated, locally advanced, unresectable or metastatic (Stage IV) programmed death-ligand 1 (PD-L1)-positive triple-negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced unresectable, histologically documented triple-negative breast cancer (TNBC) (absence of HER2-over-expression, ER, and PgR expression by local assessment)
* HER2-low-status
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* If metastatic disease (Stage IV), measurable disease outside of the bone
* No prior systemic therapy for metastatic or locally advanced unresectable TNBC
* Tumor PD-L1 expression as documented through central testing of a representative tumor tissue specimen
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate hematologic and end-organ function
* Negative HIV test at screening, with the following exception: individuals with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200/uL, and have an undetectable viral load
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Positive hepatitis B surface antibody (HBsAb) test at screening, or a negative HBsAb at screening accompanied by either of the following: negative hepatitis B core antibody (HBcAb); positive HBcAb test followed by quantitative hepatitis B virus (HBV) DNA < 500 IU/mL
* Negative hepatitis C virus (HCV) antibody test at screening, or a positive HCV antibody test followed by a negative HCV RNA test at screening
* Adequate cardiovascular function

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 4 months after the final dose of tobemstomig or pembrolizumab, and 6 months after the final dose of nab-paclitaxel
* Poor venous access
* History of malignancy within 5 years prior to consent, except for the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, nonmelanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Hypercalcemia or hypercalcemia that is symptomatic
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis (granulomatosis with polyangiitis), Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Active tuberculosis (TB)
* Significant cardiovascular/cerebrovascular disease within 3 months prior to consent
* History or presence of an abnormal ECG that is deemed clinically significant
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease (e.g., severe left ventricular systolic dysfunction, left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome
* Major surgical procedure within 4 weeks prior to initiation of study treatment
* Treatment with therapeutic oral or IV antimicrobials (anti-bacterial, anti-fungal, antiviral, anti-parasitic) within 1 week prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the participant at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 28 days prior to initiation of study treatment
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or anti-CTLA therapeutic antibodies or an anti-LAG3 agent
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including, but not limited to, prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents) within 2 weeks prior to initiation of study treatment
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the tobemstomig or pembrolizumab formulation
* Known allergy or hypersensitivity to any component of the to nab-paclitaxel formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 24 months)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Two consecutive occasions at least 4 weeks apart (up to approximately 24 months)
Duration of Response (DOR) | From the first occurrence of a confirmed objective response to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 24 months)
Overall Survival (OS) | From randomization to death from any cause (up to approximately 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (5):
  - Cancer Blood and Specialty Clinic, Los Alamitos, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Novant Health Presbyterain Medical Center, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
- Centro de Investigaciones Médicas y Desarrollo LC S.R.L, Buenos Aires, Argentina
- Sunshine Hospital, St Albans, Victoria, Australia
- Brazil (4):
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
- Fakultni Thomayerova nemocnice, Praha 4 - Krc, Czechia
- Germany (3):
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH, Essen
  - Dres. Andreas Köhler und Roswitha Fuchs, Langen
  - Universitätsklinikum Ulm Am Michelsberg, Ulm
- Komarom-Eszergom Varmegyei Szent Borbala Korhaz, Tatabánya, Hungary
- Israel (2):
  - Hadassah University Hospital - Ein Kerem, Jerusaelm
  - Sheba Medical Center, Ramat Gan
- Italy (2):
  - Ospedale Provinciale Santa Maria Delle Croci, Ravenna, Emilia-Romagna
  - Ospedale San Raffaele, Milan, Lombardy
- Mexico (4):
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - OncoMed, Mexico City, Mexico CITY (federal District)
  - Centro Médico Zambrano Hellion, Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
- Peru (4):
  - Centro Medico Monte Carmelo, Arequipa
  - Oncosalud Sac, Lima
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Instituto Peruano de Oncología y Radioterapia, Lima
- Poland (2):
  - ?wi?tokrzyskie Centrum Onkologii, Kielce
  - Szpital Uniwersytecki w Krakowie, Oddzia? Kliniczny Kliniki Onkologii, Krakow
- Medical Oncology Centre of Rosebank, Johannesburg, South Africa
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (2):
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
- National Taiwan Uni Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing